CLINICAL TRIAL: NCT01551589
Title: Multicenter Prospective Randomized Phase III Trial Comparing Elective to Prophylactic Regional Lymph Node Irradiation for Thoracic Esophageal Cancer
Brief Title: Involved Field Irradiation (IFI) Versus Elective Nodal Irradiation (ENI) for Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengya Chou (Other)
Responsible Party: Sponsor-Investigator, Chengya Chou, Chairman of Radiotherapy department, The Second People's Hospital of Sichuan
Organization: The Second People's Hospital of Sichuan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSWOG0001; BT-IST-SCCHN-037 (Other: BT-IST-SCCHN-037)
Record Dates: First submitted 2012-03-04; First posted 2012-03-13 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; Concurrent chemoradiotherapy; Clinical target volume; Safety; Prognosis
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Involved Field Irradiation(IFI) (Experimental): Involved Field Irradiation(IFI):The clinical target volume of regional lymph node (CTVn) of IFI included the nodal region(s) in which the involved lymph node(s) was/were located.chemothrapy:docetaxel and cisplatin.
  Interventions: Radiation: Involved Field Irradiation(IFI); Drug: docetaxel and cisplatin
- Elective Nodal Irradiation (ENI) (Active Comparator): Elective Nodal Irradiation (ENI):The CTVn of ENI included the involved lymph node regions and clinically uninvolved lymph nodal stations according to the location of primary tumor. Lymph node station numbers 1/2/4/5/7, 2/4/5/7 and 4/5/7/16/17 were included for upper, middle and lower thoracic ESCC in the ENI arm respectively.chemothrapy:docetaxel and cisplatin.
  Interventions: Drug: docetaxel and cisplatin; Radiation: Elective Nodal Irradiation (ENI)

INTERVENTIONS:
Radiation: Involved Field Irradiation(IFI) — Involved Field Irradiation(IFI):only irradiate positive lymph node by CT or PET-CT Radiation: IMRT IMRT is administered with chemotherapy from week 1 to week 8PTV-GTV（primary tumor）：66-70Gy/33~35F，once a day, 5 times per week PTV-CTV（Clinical target,primary tumor extended 3cm in Axial）：50-56Gy/33~35f，once a day, 5 times per week PTV-GTVnd（positive node）：66-70Gy/33~35F，once a day, 5 times per week.
  Arms: Involved Field Irradiation(IFI)
Drug: docetaxel and cisplatin — Drug: docetaxel and cisplatin.Consists of docetaxel 60-80mg/m2 day 1 and cisplatin 25mg/m2 days 1 to 3, repeat every 3 weeks, for 2 cycles.
  Other Names: chemothrrapy
Radiation: Elective Nodal Irradiation (ENI) — The CTVn of ENI included the involved lymph node regions and clinically uninvolved lymph nodal stations according to the location of primary tumor. Lymph node station numbers 1/2/4/5/7, 2/4/5/7 and 4/5/7/16/17were included for upper, middle and lower thoracic ESCC in the ENI arm respectively.
  Arms: Elective Nodal Irradiation (ENI)

SUMMARY:
This study examines contrast advantages and disadvantages of elective or prophylactic nodal irradiation in the treatment of esophageal cancer with three-dimensional conformed radiotherapy.

DETAILED DESCRIPTION:
Esophageal lymph node drainage area is rich, according to different sites, easy to metastasis to different regions. For patient underwent concurrent chemoradiotherapy, how reasonable design the clinical target volume of lymph node drainage area has always been controversial, one is to irradiate positive lymph nodes only, the other is to irradiate the easier involved lymph node area according to different sites, in order to contrast advantages and disadvantages of the two kind of target area design，so the study was designed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80
2. ECOG performance status 0-2
3. Weight is not less than 90% of it before treatment
4. Histologically proven primary thoracic esophageal squamous cell carcinoma previously untreated stage I-III
5. Chest and abdominal contrast enhanced CT within 2 weeks prior to registration(PET/CT scan is selective)
6. WBC ≥ 4.0X109/L ,Absolute neutrophil count (ANC) ≥ 2.0X109/L
7. Platelets ≥ 100X109/L
8. Hemoglobin ≥ 90g/L(without blood transfusion)
9. AST (SGOT)/ALT (SGPT) ≤ 2.5 x upper limit of normal, Bilirubin ≤ 1.5 x upper limit of normal
10. Creatinine ≤ 1.5 x upper limit of normal
11. Sign study-specific informed consent prior to study entry -

Exclusion Criteria:

1. Multiple primary esophageal tumors
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
3. Severe, active comorbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months
   * Transmural myocardial infarction within the last 6 months
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   * Acquired immune deficiency syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
4. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
5. Prior systemic chemotherapy, prior radiation therapy or prior target drug therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
radiation pneumonitis and radiation esophagitis | Acute and late toxicities of lung and esophagus were evaluated according to RTOG criteria with CT scans every 3 months for 1 years
  radiation pneumonitis and radiation esophagitis,

SECONDARY OUTCOMES:
3-year Overall survival(OS) | CT scans performed every 6 months for 3 years
  3-year Overall survival(OS)
3-year Disease-free survival | CT scans every 6 months for 3 years
  3-year Disease-free survival
Quality of life(QoL) | Evaluation of quality of life every week for 3 months
  Quality of life(QoL)
Local control rate/ Inside irrational field recurrence rate | 2 year
  Evaluation after treatment 3 months and two years in the tumor local control and key observation radiation fields inside and outside the tumor recurrence and lymph node metastatic rate. To guide the rational clinical target volume of lymph node of esophageal cancer underwnet concurrent chemoradiotherapy and to Prolong the survival time, improve the quality of life of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: JINYI LANG, M.D., Study Chair — The Second People's Hospital of Sichuan
Locations (4):
- China (4):
  - Guangxi Tumor Hospital, Nanning, Guangxi
  - GuiZhou Cancer Hospital, Guiyang, Guizhou
  - The Second People's Hospital of Sichuan, Chengdu, Sichuan
  - Yunnan Tumor Hospital, The Third Affiliated Hospital of KUNMING Medical University, Kunming, Yunnan